CLINICAL TRIAL: NCT00424541
Title: A Multiple Center, Randomized, Double Blind, Parallel Group, Multiple Oral Doses Study to Evaluate the Pharmacokinetic and Pharmacodynamic Profiles of 150 mg and 300 mg of SPP100 in Japanese Patients With Mild to Moderate Essential Hypertension
Brief Title: Pharmacokinetic and Pharmacodynamic Profiles of Aliskiren in Japanese Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A1104
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2007-11

CONDITIONS: Hypertension
Keywords: Pharmacokinetics, pharmacodynamics, safety, RAS profile, SPP100, aliskiren, Japanese, essential hypertension; Mild to moderate essential hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: SPP100 (aliskiren)

SUMMARY:
This study will evaluate the pharmacokinetic profile, the effect of rennin inhibition and the relationship among pharmacokinetics, renin-angiotensin system (RAS) biomarkers, and blood pressure lowering effects of oral doses of SPP100 in Japanese patients with mild to moderate essential hypertension. Safety will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with mild to moderate essential hypertension aged 20 to 80 years
* Blood pressure: Mean (based on 3 recordings at 1-2 minute intervals) sitting diastolic blood pressure values on 14 days or 3 days before the treatment should meet the following criteria:

  * 14 days before treatment: ≥ 90 mmHg and < 110 mmHg
  * 3 days before treatment: ≥ 95 mmHg and < 110 mmHg
  * The difference in mean sitting diastolic blood pressure between 14 days and 3 days before the treatment is within 10 mmHg
* Body weight no less than 50 kg

Exclusion Criteria:

* Patients with mean (based on 3 recordings at 1-2 minute intervals) systolic blood pressure ≥ 180 mmHg and/or mean diastolic blood pressure ≥ 110 mmHg at Day -28, Day -14 and Day -3.
* Patients with or suspected of having secondary hypertension
* Patients suspected of having malignant hypertension

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2007-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic profile of aliskiren administration after meal Day 1, Day 14, and Day 28

SECONDARY OUTCOMES:
effect of aliskiren on the RAS profile
relationship among steady state pharmacokinetics, change in RAS biomarkers and blood pressure lowering effect of aliskiren
safety

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative Site
Locations (1):
- Novartis Investigative Site, Tokyo, Japan

REFERENCES:
- See also: Results for CSPP100A1104 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2500